CLINICAL TRIAL: NCT00961025
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single/Multiple Dosing, Dose Escalation Clinical Phase 1 Study to Investigate the Safety, Tolerance, and Pharmacokinetics/Pharmacodynamics of DA-1229 in Healthy Male Subjects
Brief Title: A Study to Characterize the Pharmacokinetics/Pharmacodynamics and Effect of Food of DA-1229 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: KEUMJAE KO / Assistant Manager, Clinical Development Team 1
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA1229_DM_I
Record Dates: First submitted 2009-08-10; First posted 2009-08-18 (Estimated); Last update posted 2009-08-24 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitis Type 2
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DA-1229 (Experimental): DA-1229
  Interventions: Drug: DA-1229

INTERVENTIONS:
Drug: DA-1229 — single dose study : DA-1229 1.25,2.5,5,10,20,40,60mg
  multiple dose study : DA-1229 5,10,20,40mg
  Arms: DA-1229
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
This is a dose block-randomized, double-blind, placebo-controlled, single/multiple dosing, dose-escalation study. The study is designed to describe the relationship between multiple doses and pharmacokinetic/pharmacodynamic parameters of DA-1229 as well as safety profile.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years healthy male subjects
* Body weight :50-90kg, BMI between 18.5-25
* Blood glucose level of 70-110mg/dL on the FPG test

Exclusion Criteria:

* have a family history of diabetes
* Serum AST(SGOT), ALT(SGPT)>1.25 times upper limit of normal
* Creatinine clearance rate<80mL/min
* show SBP =<100mmHg or >=150mmHg, or DBP=<65mmHg or >=95mmHg, or tachycardia (PR>=100times/min)
* have a history of drug abuse or show positive for drug abuse or cotinine at urine screening
* smokers
* can not digest high-fat or high-calorie food(applicable only for the 10mg dose group subjects

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To characterize the pharmacokinetic/pharmacodynamic of DA-1229 in healthy male subjects | Multiple blood and urine samples will be collected for 120 hours after dosing of DA-1229

SECONDARY OUTCOMES:
To evaluate the safety and tolerance of DA-1229 | up to 10 days (single dose study), 17 days (single dose study for food effect), 20 days (multiple dose study)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, Chongo-Gu, Yon-Gon Dong, South Korea

REFERENCES:
- [Derived] Kim TE, Lim KS, Park MK, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. Evaluation of the pharmacokinetics, food effect, pharmacodynamics, and tolerability of DA-1229, a dipeptidyl peptidase IV inhibitor, in healthy volunteers: first-in-human study. Clin Ther. 2012 Sep;34(9):1986-98. doi: 10.1016/j.clinthera.2012.08.006. Epub 2012 Sep 1. PMID 22943970